CLINICAL TRIAL: NCT02229214
Title: A Phase IV, Single-Center, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Effect of VI-0521 on the Glomerular Filtration Rate of Healthy Overweight or Obese Subjects
Brief Title: Effect of VI-0521 (Qsymia®) on Glomerular Filtration Rate (GFR) in Overweight or Obese Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OB-404
Record Dates: First submitted 2014-08-26; First posted 2014-09-01 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: Renal function; Glomerular Filtration Rate; Kidney function; Qsymia; Iohexol; Serum Creatinine; Creatinine clearance; Renal Clearance; VI-0521; Healthy volunteers
MeSH Terms: conditions — Obesity | interventions — Qsymia; Phentermine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VI-0521 (Qsymia) (Experimental): * Days 1-3: VI-0521 (Phentermine/Topiramate 3.75 mg/23 mg)
  * Days 4-6: VI-0521 (Phentermine/Topiramate 7.5 mg/46 mg)
  * Days 7-9: VI-0521 (Phentermine/Topiramate 11.25 mg/69 mg)
  * Days 10-28: VI-0521 (Phentermine/Topiramate 15 mg/92 mg)
  Interventions: Drug: Qsymia
- Sugar pill (Placebo Comparator): Days 1-28: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qsymia
  Other Names: VI-0521; Phentermine and Topiramate ER (Extended Release)
  Arms: VI-0521 (Qsymia)
Drug: Placebo
  Other Names: Sugar Pill
  Arms: Sugar pill

SUMMARY:
The main purpose of this study is measure the effect of VI-0521 on kidney function. Specifically, glomerular filtration rate (GFR) will be measured at baseline, after 4 weeks of study treatment, and after an additional 4 weeks of off-treatment recovery.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single-site study in healthy overweight or obese male and female volunteers. Oral VI-0521 (combination of phentermine and topiramate [PHEN/TPM] extended-release capsule) will be administered daily as follows:

* Days 1-3: PHEN/TPM 3.75 mg /23 mg
* Days 4-6: PHEN/TPM 7.5 mg /46 mg
* Days 7-9: PHEN/TPM 11.25 mg /69 mg
* Days 10-28: PHEN/TPM 15 mg /92 mg

A single dose of Iohexol (a non-radioactive iodine-containing contrast agent) will be administered intravenously on three separate occasions.

The study will include a total of 50 healthy subjects (40 active and 10 placebo), all of whom will have overnight stays on 3 separate occasions.

Total study duration is approximately 10 weeks (2 weeks screening, 4 weeks study treatment, 4 weeks post treatment follow up).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female 18 - 65 years of age, medically healthy with no clinically significant screening abnormalities
* BMI of ≥27 to ≤45 kg/m2
* No use of any medication (prescription, over the counter (OTC) or herbal preparations) with the exception of contraception for the entirety of the study

Key Exclusion Criteria:

* Allergy or hypersensitivity to radio contrast media, iodine or shellfish
* Plans to significantly alter their diet through fasting, very low caloric intake, elimination of certain foods (gluten, milk, meat, etc.) or similar
* Plans to undertake a significant change to physical exercise levels (i.e., initiate training for a marathon) during the study period
* Consumption of a high protein diet or protein/body building meal supplementation and/or replacement. The use of any product containing creatine is strictly prohibited
* History of glaucoma or increased intraocular pressure
* History of bipolar disorder or psychosis, history of psychiatric hospitalization, greater than one lifetime episode of major depression, current depression of moderate or greater severity, presence or history of suicidal behavior or ideation with some intent to act on it
* Cholelithiasis (gallstones) within the past 6 months
* History of nephrolithiasis (kidney stones)
* Evidence of any clinically significant renal, pulmonary, hepatic, psychiatric or other condition by history, physical examination or laboratory studies that, in the opinion of the investigator, would contraindicate the administration of study medications, affect compliance, interfere with study evaluations or confound the interpretation of study results as determined by the investigator
* Current use of any tobacco products including cigarettes, cigars, pipes, and chewing tobacco, or nicotine replacement products (e.g., patch, gum, lozenge, etc.), or chronic use within the previous three months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Galloway, MD, Principal Investigator
Locations (1):
- Research Center, Lakewood, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- VI-0521 (Qsymia): * Days 1-3: VI-0521 (Phentermine/Topiramate 3.75 mg/23 mg)
  * Days 4-6: VI-0521 (Phentermine/Topiramate 7.5 mg/46 mg)
  * Days 7-9: VI-0521 (Phentermine/Topiramate 11.25 mg/69 mg)
  * Days 10-28: VI-0521 (Phentermine/Topiramate 15 mg/92 mg)
  Qsymia
- Placebo: Days 1-28: Placebo
  Sugar Pill
Period: Overall Study
Arm/Group | VI-0521 (Qsymia) | Placebo
Started | 41 | 10
Completed | 35 | 10
Not Completed | 6 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Days 1-28: Placebo
  Placebo (sugar pill)
- Total: Total of all reporting groups
Arm/Group | VI-0521 (Qsymia) | Placebo | Total
Number analyzed (Participants) | 41 | 10 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.4 (11.07) | 37.6 (9.80) | 38.2 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 4 | 31
  Male | 14 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 3 | 16
  Not Hispanic or Latino | 28 | 7 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 30 | 8 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 41 | 10 | 51
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 33.2 (4.72) | 31.3 (2.81) | 32.8 (4.46)
iGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 95.1 (14.05) | 87.3 (9.06) | 93.6 (13.49)

OUTCOME MEASURES:

1. Primary Outcome: Change in iGFR (Glomerular Filtration Rate as Measured by Iohexol Clearance) From Baseline to End of Treatment
Description: Method that uses iohexol clearance and body surface area to measure kidney function.
  Iohexol is an FDA-approved non-radioactive iodine-containing substance widely used in radio-imaging procedures and as a marker for the measurement of in GFR.
Time Frame: Baseline, end of treatment
Population: The number analyzed in this outcome measure are those subjects who have both baseline and end of treatment iGFR measurements.
Measure: Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | VI-0521 (Qsymia) | Placebo
Number analyzed (Participants) | 34 | 10
mL/min/1.73 m^2 | -14.92 (1.28) | 1.08 (2.28)

2. Secondary Outcome: Change in Serum Creatinine From Baseline to End of Treatment
Time Frame: Baseline, end of treatment
Population: The number analyzed in this outcome measure are those subjects who have both baseline and end of treatment serum creatininine measurements
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Sugar Pill: Days 1-28: Placebo
  Placebo
Arm/Group | VI-0521 (Qsymia) | Sugar Pill
Number analyzed (Participants) | 35 | 10
mg/dL | 0.10 (0.01) | 0.03 (0.03)

3. Secondary Outcome: Change in Serum Creatinine From Baseline to 28 Days After End of Treatment
Time Frame: Baseline, 28 days after end of treatment
Population: The number analyzed in this outcome measure are those subjects who have both baseline and 28 days after end of treatment serum creatinine measurements.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | VI-0521 (Qsymia) | Sugar Pill
Number analyzed (Participants) | 35 | 10
mg/dL | -0.01 (0.01) | 0.03 (0.02)

4. Secondary Outcome: Change in Cystatin C From Baseline to End of Treatment
Time Frame: Baseline, end of treatment
Population: The number analyzed in this outcome measure are those subjects who have both baseline and end of treatment cystatin C measurements.
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | VI-0521 (Qsymia) | Placebo
Number analyzed (Participants) | 35 | 10
mg/L | 0.04 (0.01) | 0.03 (0.02)

5. Primary Outcome: Change in iGFR (Glomerular Filtration Rate as Measured by Iohexol Clearance) From Baseline to 28 Days After End of Treatment
Description: as for outcome 1
Time Frame: Baseline, 28 days after end of treatment
Population: The number analyzed in this outcome measure are those subjects who have both baseline and 28 days after treatment iGFR measurements.
Measure: Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | VI-0521 (Qsymia) | Sugar Pill
Number analyzed (Participants) | 32 | 10
mL/min/1.73 m^2 | -3.75 (1.49) | 2.34 (1.34)

6. Secondary Outcome: Change in Cystatin C From Baseline to 28 Days After End of Treatment
Time Frame: Baseline, 28 days after end of treatment
Population: The number analyzed in this outcome measure are those subjects who have both baseline and 28 days after end of treatment cystatin C measurements.
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | VI-0521 (Qsymia) | Placebo
Number analyzed (Participants) | 35 | 10
mg/L | 0.01 (0.01) | 0.02 (0.01)

7. Secondary Outcome: Percentage of Subjects With a Decrease of >/= 15% in Iohexol Clearance From Baseline to End of Treatment
Time Frame: Baseline, end of treatment
Measure: Number; unit: percent of participants
Arm/Group | VI-0521 (Qsymia) | Placebo
Number analyzed (Participants) | 41 | 10
percent of participants | 48.8 | 0

8. Secondary Outcome: Percentage of Subjects With a Decrease of >/= 15% in Iohexol Clearance From Baseline to 28 Days After End of Treatment
Time Frame: Baseline, 28 days after end of treatment
Measure: Number; unit: percent of participants
Arm/Group | VI-0521 (Qsymia) | Placebo
Number analyzed (Participants) | 41 | 10
percent of participants | 7.3 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | VI-0521 (Qsymia) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/10
Other Adverse Events (participants affected / at risk) | 33/41 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VI-0521 (Qsymia) (N=41) | Placebo (N=10)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Subject was inside a boom trimming trees when the middle of the metal arm of the boom broke and resulted in subject falling.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VI-0521 (Qsymia) (N=41) | Placebo (N=10)
Ocular Hyperaemia (Eye disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Paraesthesia Oral (Gastrointestinal disorders) | 3 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 12 | 0
Headache (Nervous system disorders) | 9 | 2
Dizziness (Nervous system disorders) | 7 | 0
Insomnia (Psychiatric disorders) | 5 | 0
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days